CLINICAL TRIAL: NCT00002521
Title: HIGH-DOSE CYCLOPHOSPHAMIDE, ETOPOSIDE, AND CISPLATIN (CEP) WITH RESCUE BY AUTOLOGOUS BONE MARROW OR AUTOLOGOUS PERIPHERAL BLOOD STEM CELLS IN PATIENTS WITH RELAPSED OR REFRACTORY NON-HODGKIN'S LYMPHOMA (INTERMEDIATE AND HIGH-GRADE HISTOLOGIES)
Brief Title: Combination Chemotherapy and Bone Marrow and/or Peripheral Stem Cell Transplantation in Treating Patients With Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Temple University (Other)
Responsible Party: Temple University Bone Marrow Transplant Program, Temple Univeristy Health Systems
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000078282; TUHSC-2161; NCI-V93-0248
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2010-10-01 (Estimated); Status verified 2010-09

CONDITIONS: Lymphoma
Keywords: stage I adult diffuse small cleaved cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I adult Burkitt lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult lymphoblastic lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma | interventions — Cisplatin; Cyclophosphamide; Etoposide; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: cyclophosphamide
Drug: etoposide
Procedure: autologous bone marrow transplantation
Procedure: bone marrow ablation with stem cell support
Procedure: peripheral blood stem cell transplantation
Procedure: syngeneic bone marrow transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Bone marrow and peripheral stem cell transplantation may allow doctors to give high doses of chemotherapy and kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy with cyclophosphamide, etoposide and cisplatin followed by bone marrow and/or peripheral stem cell transplantation in patients with relapsed or refractory intermediate- or high-grade non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the curative potential of high-dose cyclophosphamide, etoposide, and cisplatin (CEP) with syngeneic or autologous bone marrow and/or autologous peripheral blood stem cell rescue in patients with relapsed or refractory, stage I-IV, intermediate- or high-grade non-Hodgkin's lymphoma.
* Determine the overall response rate and survival of patients treated with this regimen.
* Determine the toxic effects of this regimen in these patients.
* Determine the differences in the rates of engraftment, response, and survival of patients treated with bone marrow vs peripheral blood stem cell transplantation.
* Determine the response rate and survival of patients treated with consolidative radiotherapy after recovery from transplantation.
* Determine the toxic effects of consolidative radiotherapy after recovery from transplantation in these patients.

OUTLINE: Syngeneic or autologous bone marrow and/or autologous peripheral blood stem cells (PBSC) are harvested. Syngeneic bone marrow transplantation is preferred for patients with a qualifying identical twin donor. Patients without a syngeneic donor who have a history of lymphomatous involvement of the bone marrow and are profoundly hypocellular undergo harvest of PBSC alone. Patients without a syngeneic donor who have no history of lymphomatous involvement of the bone marrow undergo harvest of autologous bone marrow or PBSC.

Patients receive conditioning comprising cyclophosphamide IV over 1 hour on days -6 to -3 and etoposide IV over 1 hour every 12 hours and cisplatin IV continuously on days -6 to -4. Bone marrow and/or PBSC are infused on day 0. (Patients requiring more than 25 bags of stem cells receive bone marrow transplantation on day 0 and PBSC transplantation on day 1.)

After recovery from transplantation, eligible patients receive consolidative radiotherapy to any site of prior bulk disease (greater than 5 cm) present at any time before transplantation and any site of disease present at the time of transplantation.

Patients are followed at 3, 6, and 12 months and then annually thereafter.

PROJECTED ACCRUAL: A maximum of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven relapsed or refractory, stage I-IV, intermediate- or high-grade non-Hodgkin's lymphoma

  * Eligible subtypes:

    * Diffuse small cleaved cell
    * Diffuse mixed (small and large cell)
    * Diffuse large cell
    * Large cell immunoblastic
    * Lymphoblastic
    * Small noncleaved cell
* High-grade histology patients should first be considered for Protocol TUHSC-1520
* Must have chemosensitive disease, defined by 1 of the following conditions:

  * Response to initial chemotherapy without obtaining complete response (CR)(refractory lymphoma)
  * Relapse after chemotherapy-induced CR if tumor volume reduced by at least 25% for more than 1 month after completion of 1-3 courses of salvage chemotherapy (chemosensitive relapse)
* No chemoresistant disease, defined by the following conditions:

  * Unresponsive or progressive disease during initial chemotherapy
  * Relapse after chemotherapy-induced CR if tumor volume not reduced by at least 25% after completion of 1-3 courses salvage chemotherapy (chemoresistant relapse)
* No CNS involvement by lymphoma
* Syngeneic bone marrow transplantation offered to patients with consenting identical twin donor NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age:

* 15 to 60 (physically fit patients up to age 70 may be considered)

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* AST and ALT not persistently greater than 2 times normal

Renal:

* Creatinine less than 1.8 mg/dL

Cardiovascular:

* Cardiac ejection fraction at least 45%

Pulmonary:

* DLCO, FEV_1, and FVC at least 50% predicted
* Resting pO_2 at least 70 mm Hg

Other:

* HIV negative
* No other concurrent disease that would limit life expectancy
* No active infection
* No severe neurologic or emotional disorders
* Not pregnant
* Fertile patients must use effective contraception
* Adequate psychological support available

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1993-02; Primary Completion 2000-02 (Actual); Study Completion 2000-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth F. Mangan, MD, FACP, Study Chair — Fox Chase Cancer Center
Locations (1):
- Fox Chase - Temple Cancer Center, Philadelphia, Pennsylvania, United States